CLINICAL TRIAL: NCT00206843
Title: Rapid Emergency Department Heart Failure Outpatient Trial (REDHOT II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 005
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Results available (Experimental)
  Interventions: Device: Triage BNP Test
- Results blinded (No Intervention)

INTERVENTIONS:
Device: Triage BNP Test
  Arms: Results available

SUMMARY:
The purpose of this study is to test whether physicians can make more informed treatment, admission, and discharge decisions related to patient care by having serial Triage® BNP test results available to assess disease severity, while patients are being treated for HF in the Emergency Department and/or during their admission. This is believed to lead to a better outcome as well as more efficient and cost-effective treatment.

DETAILED DESCRIPTION:
This is a patient-randomized clinical study consisting of patients who present to the ED requiring treatment and/or admission for HF. At each site, patients will be randomized into either a control arm or an experimental arm. Serial blood samples will be collected from all patients throughout their stay in the ED and the hospital. In the experimental arm, the Triage® BNP test will be performed on all blood samples collected and each BNP result will be made available to the attending physicians immediately. In the control arm, blood samples will not be analyzed on-site for BNP but instead sent directly to Biosite Inc. for testing.A comparison will be made between the control and experimental arms of the study to determine if there are any significant differences in length of stay, re-hospitalizations, all cause mortality, BNP levels, quality of life, and costs to treat patients.

ELIGIBILITY:
Inclusion Criteria:

Age 18 and older Patient needs treatment for HF

Exclusion Criteria:

Current MI or ACS with ST deviation of 1 mm or greater Renal failure requiring dialysis Undergone hemodialysis within the last month Enrollment (Baseline) Triage® BNP concentration = 100 pg/ml or less Enrolled in any other drug trial or receiving an experimental treatment for HF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2004-11; Primary Completion 2007-04 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay
Combined cardiac related re-hospitalizations and all cause mortality (14-day and 30-day)

SECONDARY OUTCOMES:
Discharge BNP
Change in BNP from enrollment to discharge (ΔBNP)
Ratio of ΔBNP/length of stay
Cost Effectiveness
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Judd E Hollander, MD, Principal Investigator — University of Pennsylvania
Locations (10):
- United States (10):
  - Chandler Regional Hospital, Chandler, Arizona
  - University of California, San Diego MedicalCenter, San Diego, California
  - Detroit Receiving Hospital/Wayne State University, Detroit, Michigan
  - Sinai Grace Hospital/Wayne State, Detroit, Michigan
  - Beaumont Hospital, Troy, Troy, Michigan
  - New York Methodist Hospital, Brooklyn, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania